CLINICAL TRIAL: NCT06009926
Title: Phase II Randomized, Double-Blind, Placebo-Controlled Trial of Broccoli Seed and Sprout Extract (BSSE) to Evaluate Detoxification of Carcinogens in Firefighters
Brief Title: Evaluation of Broccoli Seed and Sprout Extract for Detoxification of Carcinogens in Firefighters
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2023-06404; NCI-2023-06404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00003544 (Other: University of Arizona Cancer Center - Prevention Research Clinic); UAZ22-11-01 (Other: DCP); P30CA023074 (NIH); UG1CA242596 (NIH)
Record Dates: First submitted 2023-08-23; First posted 2023-08-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm; Occupational Malignant Neoplasm
MeSH Terms: interventions — Acetaminophen; Specimen Handling; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigators and clinical research coordinators will avoid speculating with the participant regarding the participant's treatment group. The individual authorized to break the blind, if conditions are met, is the study principal investigator in consultation with the Division of Cancer Prevention medical monitor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I (BSSE-placebo) (Experimental): Participants receive BSSE PO QD for 7-10 days then undergo the first flashover training between day 7-10 of agent intervention. Participants then receive placebo PO QD for 7-10 days then undergo second flashover training after a washout period of 2 weeks to 3 months. Participants also undergo urine sample collection throughout the study. (CLOSED TO ACCRUAL 10/07/2024)
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: Broccoli Sprout/Broccoli Seed Extract Supplement; Drug: Placebo Administration; Other: Questionnaire Administration; Other: Training
- Group II (placebo-BSSE) (Experimental): Participants receive placebo PO QD for 7-10 days then undergo the first flashover training between day 7-10 of agent intervention. Participants then receive BSSE for 7-10 days then undergo second flashover training after a washout period of 2 weeks to 3 months. Participants also undergo urine sample collection throughout the study. (CLOSED TO ACCRUAL 10/07/2024)
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: Broccoli Sprout/Broccoli Seed Extract Supplement; Drug: Placebo Administration; Other: Questionnaire Administration; Other: Training
- Group III (BSSE, acetaminophen) (Experimental): Participants receive BSSE PO QD for 12 weeks on study. Participants also receive acetaminophen PO once prior to starting BSSE and once following completion of BSSE on study. Participants undergo blood and urine sample collection throughout the study.
  Interventions: Drug: Acetaminophen; Procedure: Biospecimen Collection; Dietary Supplement: Broccoli Sprout/Broccoli Seed Extract Supplement; Other: Questionnaire Administration
- Group IV (placebo, acetaminophen) (Active Comparator): Participants receive placebo PO QD for 12 weeks on study. Participants also receive acetaminophen PO once prior to starting placebo and once following completion of placebo on study. Participants undergo blood and urine sample collection throughout the study.
  Interventions: Drug: Acetaminophen; Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Acetaminophen — Given PO
  Other Names: APAP; Paracetamol; Tylenol
  Arms: Group III (BSSE, acetaminophen); Group IV (placebo, acetaminophen)
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Dietary Supplement: Broccoli Sprout/Broccoli Seed Extract Supplement — Given PO
  Other Names: Avmacol
  Arms: Group I (BSSE-placebo); Group II (placebo-BSSE); Group III (BSSE, acetaminophen)
Drug: Placebo Administration — Given PO
  Arms: Group I (BSSE-placebo); Group II (placebo-BSSE); Group IV (placebo, acetaminophen)
Other: Questionnaire Administration — Ancillary studies
Other: Training — Undergo flashover training
  Other Names: Training Programs
  Arms: Group I (BSSE-placebo); Group II (placebo-BSSE)

SUMMARY:
This phase II randomized, placebo-controlled trial evaluates whether daily supplementation with broccoli seed and sprout extract (BSSE), also known as Avmacol Extra Strength (ES), enhances the body's natural ability to detoxify carcinogens commonly encountered by firefighters. Firefighters are routinely exposed to harmful chemicals such as benzene and polycyclic aromatic hydrocarbons (PAHs) through smoke inhalation, structural fires, and fuel leak incidents exposures that contribute to their elevated cancer risk. BSSE contains bioactive compounds known to activate phase II detoxification enzymes that help eliminate reactive toxins from the body. A single dose of acetaminophen (Tylenol) is administered at both baseline and end-of-intervention as a metabolic probe to assess changes in detoxification enzyme activity. Acetaminophen is metabolized through the same pathways as benzene and PAHs, making it a useful surrogate for evaluating the effect of BSSE on the detoxification of fire-related toxicants. Participants were originally randomized into one of total four study groups. Groups I and II, now closed to accrual, were designed to assess BSSE effects before and after controlled flashover fire training exercises. These arms were discontinued after it was determined that training fires produced insufficient real-world toxicant exposure to evaluate the intervention's impact. Groups III and IV were subsequently open and represent the active phase of the study. Group III participants receive BSSE daily for 12 weeks, while Group IV participants receive a matched placebo. Both groups include acetaminophen challenge at baseline and end-of-intervention, with biospecimen collection to evaluate detoxification capacity and explore genetic and epigenetic modifiers of response. Although the protocol includes four study groups, only two are currently active. Groups I and II remain part of the study record but are closed and will not contribute to the primary outcome analyses.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether BSSE increases the urinary excretion of mercapturic acid of acetaminophen, a surrogate for detoxification of the carcinogen benzene in healthy, incumbent firefighters.

SECONDARY OBJECTIVES:

I. To evaluate the effects of BSSE on urinary excretion of acetaminophen glucuronide, a surrogate for detoxification of polycyclic aromatic hydrocarbons (PAHs).

II. To evaluate the safety and tolerability of BSSE.

EXPLORATORY OBJECTIVES:

I. To determine whether the GSTM1 and GSTT1 genotypes are important genetic modulators of BSSE-induced detoxification of carcinogens.

II. To evaluate the effects of BSSE on urinary metabolomics. III. To determine the effects of BSSE on the urinary excretion of the mercapturic acid of benzene after fire/fuel leak activities.

IV. To determine the effects of BSSE on the urinary excretion of metabolites of PAHs after fire/fuel leak activities.

V. To determine the effects of BSSE on epigenetic modifications (blood microribonucleic acid [RNA] and deoxyribonucleic acid [DNA] methylation).

OUTLINE: Participants are randomized to Group III or Group IV.

GROUP I (BSSE-PLACEBO) (CLOSED TO ACCRUAL 10/07/2024): Participants receive BSSE orally (PO) daily (QD) for 7-10 days then undergo the first flashover training between day 7-10 of agent intervention. Participants then receive placebo PO QD for 7-10 days then undergo second flashover training after a washout period of 2 weeks to 3 months. Participants also undergo urine sample collection throughout the study.

GROUP II (PLACEBO-BSSE) (CLOSED TO ACCRUAL 10/07/2024): Participants receive placebo PO QD for 7-10 days then undergo the first flashover training between day 7-10 of agent intervention. Participants then receive BSSE for 7-10 days then undergo second flashover training after a washout period of 2 weeks to 3 months. Participants also undergo urine sample collection throughout the study.

GROUP III: Participants receive BSSE PO QD for 12 weeks on study. Participants also receive acetaminophen PO once prior to starting BSSE and once following completion of BSSE on study. Participants undergo blood and urine sample collection throughout the study.

GROUP IV: Participants receive placebo PO QD for 12 weeks on study. Participants also receive acetaminophen PO once prior to starting placebo and once following completion of placebo on study. Participants undergo blood and urine sample collection throughout the study.

After completion of study intervention, participants are followed up at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female incumbent firefighters who are current non-smokers.
* Age >= 18 years.
* Karnofsky performance scale >= 70%.
* Absolute neutrophil count >= 1,000/microliter.
* Platelets >= 100,000/microliter.
* Total bilirubin =< 2 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase [SGPT]) =< 2 x ULN.
* Creatinine =< 1.5 x ULN.
* Participants on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible.
* The effects of BSSE on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of invasive cancer within the past 2 years, except for excised and cured non-melanoma skin cancer or carcinoma in situ of the cervix. Participants who continue adjuvant treatment for an index cancer occurring > 2 years ago, such as adjuvant hormonal therapy for breast cancer, are excluded. Participants who are on anti-neoplastic treatment for a chronic malignancy, such as multiple myeloma or chronic myelogenous leukemia, are excluded.
* Chronic, current or recent (within the past 2 weeks) use of systemic steroid doses equivalent to prednisone > 5 mg daily for continued use > 14 days. Use of inhaled steroids, nasal sprays, and topical creams for small body areas (< 10% body surface area) is allowed.
* Participants may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Avmacol ES (BSSE).
* Uncontrolled intercurrent illness including, but not limited to, serious ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women. Pregnant women are excluded from this study because the effects of BSSE on the developing human fetus are unknown. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with BSSE, breastfeeding should be discontinued if the mother is treated with BSSE.
* Participants with known human immunodeficiency virus (HIV), chronic hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Participants with HIV, HBV and HCV are excluded from this study because there is no information regarding the impact of anti-viral drugs on the bioavailability of Avmacol ES. Sulforaphane (SF) is known to modulate certain phase 1 and phase 2 enzymes involved in drug metabolism. The potential for SF to alter the metabolism (either by increasing or decreasing) of antiviral therapy could have an effect on the efficacy of the pharmaceuticals to keep viral titers low and the disease under control. Since many of the drugs used in therapies of these viral infections have extensive CYP450 enzymatic impact and BSSE has its own enzymatic properties, there is concern for drug-to-drug interactions.
* Ongoing use of any supplements containing active compounds in cruciferous vegetables such as SF and glucoraphanin (GR). The use of supplements related to the study agent may confound the study endpoints. Participant will be eligible if they agree to stop the SF or GR product at least 14 days prior to the baseline visit.
* History of allergic reactions to acetaminophen or the formulation ingredients or any other contraindication to acetaminophen use.
* Unwilling or unable to refrain from the use of non-study acetaminophen (or acetaminophen containing products) for 72 hours prior to the baseline evaluation of acetaminophen metabolism and for 72 hours prior to the end-of-intervention evaluation of acetaminophen metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in total amount of acetaminophen mercapturate excreted in the urine | Baseline to end-of-intervention
  Will compare after acetaminophen dosing between broccoli seed and sprout extract (BSSE) and placebo arms. Will be quantified by liquid chromatography tandem mass spectrometry. Log-transformation will be applied to total amount of acetaminophen mercapturate before deriving the changes at the end of intervention from baseline since the total amount of acetaminophen mercapturate may be highly right skewed. Even if the total amount of acetaminophen mercapturate is not highly right skewed, log-transformation will also allow comparison of the relative percent change in total amount of acetaminophen mercapturate at the end of intervention from baseline between the BSSE and placebo groups through use of the geometric mean of total amount of acetaminophen mercapturate. Will be analyzed in participants who initiated treatment and provided both pre-study agent intervention and post-study agent intervention urine.

SECONDARY OUTCOMES:
Change in total amount of acetaminophen glucuronide excreted in the urine | Baseline to end-of-intervention
  Will compare after acetaminophen dosing between BSSE and placebo arms. Will be quantified by liquid chromatography tandem mass spectrometry.
Incidence of adverse events | Start of intervention to follow-up
  Will evaluate safety of BSSE, as measured by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5. Toxicity will be measured by adverse events (AE) classified in accordance with NCI CTCAE version 5. The frequency and associated percentage of each specific AE will be tabulated by treatment group and then compared via Fisher's exact test. All participants will be evaluable for toxicity from the time of their first dose of BSSE versus placebo. Descriptive statistics of the type and frequency of all AEs will be generated, including 95% confidence intervals.
Adherence rate | Up to 12 weeks
  Tolerability will be measured by adherence rate and will be compared between the BSSE and placebo via Fisher's exact test.

OTHER OUTCOMES:
GSTM1 and GSTT1 genotypes | Baseline to end-of-intervention
  Will assess whether the GSTM1 and GSTT1 genotypes are important genetic modulators of BSSE-induced detoxification of carcinogens in the setting of exposure to BSSE. Genomic deoxyribonucleic acid (DNA) will be isolated from circulating blood lymphocytes. GSTM1 and GSTT1 will be genotyped using standard methods. The correlation of GSTM1 and GSTT1 genotypes with detoxication of acetaminophen mercapturate/acetaminophen glucuronide will be assessed by linear regression for changes from baseline in the log-transformed acetaminophen mercapturate/acetaminophen glucuronide, in which BSSE and genotype indicators and interactions of BSSE, and genotype indicators are the covariates in the model. This will allow determination of whether the BSSE effect is significantly modulated by the genotypes.
Metabolomics | Baseline to end-of-intervention
  Will explore the effects of BSSE on urinary metabolomics on pre-acetaminophen spot urine collected at both baseline and at the end of intervention as well as spot urine collected after each fire/fuel leak activity will be analyzed. To explore the effects of BSSE on the urinary metabolome after fire/fuel leak activities, urinary metabolome will be measured at baseline, post fire exposure, and post study agent intervention. A linear mixed effects model with BSSE and post-intervention indicators and their interaction term as the covariates will be fitted to changes from baseline in each of the log-transformed metabolite levels. This model will allow comparison of the change between BSSE and placebo at post fire exposure and postintervention, respectively, as well as comparing the changes at post-intervention from post fire exposure between BSSE and placebo.
Mercapturic acid | Baseline to end-of-intervention
  Will evaluate the effects of BSSE on the urinary excretion of the mercapturic acid of benzene after fire/fuel leak activities. Will be quantified by liquid chromatography tandem mass spectrometry. To assess the effects of BSSE on the urinary excretion of mercapturic acid of benzene after fire/fuel leak activities, urine excretion of mercapturic acid of benzene will be measured at baseline, post fire exposure, and post study agent intervention. A linear mixed effects model with BSSE and post-intervention indicators and their interaction term as the covariates will be fitted to changes from baseline in the log-transformed levels of mercapturic acid of benzene. This model will allow comparison of the change between BSSE and placebo at post fire exposure and post-intervention, respectively, as well as comparing the changes at post-intervention from post fire exposure between BSSE and placebo.
Polycyclic aromatic hydrocarbons (PAHs) | Baseline to end-of-intervention
  Will assess the effects of BSSE on urinary excretion of the metabolites of PAHs after fire/fuel leak activities. Will be evaluated to assess detoxification of PAHs. PAH metabolites will be measured by liquid chromatography tandem mass spectrometry. PAH metabolites will be measured at baseline, post fire exposure, and post study agent intervention. A linear mixed effects model with BSSE and post-intervention indicators and their interaction term as the covariates will be fitted to changes from baseline in each of the log-transformed PAH metabolite levels. This model will allow the comparison of the change between BSSE and placebo at post fire exposure and post-intervention, respectively, as well as comparing the changes at postintervention from post fire exposure between BSSE and placebo.
Microribonucleic acid (microRNA) | Screening to end-of-intervention
  Will evaluate the effects of BSSE on epigenetic modifications (blood microRNA). Ribonucleic acid will be isolated from blood and microRNA expression will be measured. Two-sample t tests will be performed to compare changes in log-transformed expression levels between BSSE and placebo.
DNA methylation | Screening to end-of-intervention
  Will evaluate the effects of BSSE on epigenetic modifications (blood DNA methylation). DNA will be isolated from blood and analyzed. Two-sample t tests will be performed to compare changes in log-transformed expression levels between BSSE and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Malvi Savani, Principal Investigator — University of Arizona Cancer Center - Prevention Research Clinic
Locations (1):
- University of Arizona Cancer Center - Prevention Research Clinic, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- See also: Related Info — https://grants.nih.gov/policy/sharing.htm